CLINICAL TRIAL: NCT00768859
Title: Trastuzumab in a Neo-adjuvant Regimen for HER2+ Breast Cancer - the TRAIN Study
Acronym: TRAIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: G.S. Sonke, MD PhD, NKI-AVL
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M08TRA; 2008-000987-18 (EudraCT Number)
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Last update posted 2012-05-11 (Estimated); Status verified 2012-05

CONDITIONS: Breast Cancer; HER2 Positive
Keywords: breast cancer; HER2 positive; neo-adjuvant; trastuzumab; paclitaxel; carboplatin
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; Trastuzumab; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): paclitaxel, trastuzumab and carboplatin
  Interventions: Drug: paclitaxel, trastuzumab and carboplatin

INTERVENTIONS:
Drug: paclitaxel, trastuzumab and carboplatin — paclitaxel; 70 mg/m2 trastuzumab; 2 mg/kg (loading dose 4 mg/kg) carboplatin; AUC = 3

SUMMARY:
To determine the activity of the combination of paclitaxel, trastuzumab and carboplatin as neo-adjuvant treatment in patients with stage II or III HER2 positive breast cancer

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed infiltrating breast cancer.
* Stage II or stage III breast cancer.28 'Locally advanced breast cancer' patients are consequently eligible, including those with ipsilateral supraclavicular lymph node metastases. N1 status must have been demonstrated by either fine needle aspiration from an axillary lymph node or by a metastasis of >2 mm in diameter at sentinel node biopsy. Stage IIA patients are eligible if the tumor is >3 cm in diameter or if the tumor is between 2 and 3 cm in diameter but a breast conserving surgery is not possible.
* Overexpression and/or amplification of HER2 in an invasive component of the core biopsy, according to one of the following definitions:

  * >10% of invasive tumor cells showing strong complete circumferential membrane staining (score 3+)
  * >10% of invasive tumor cells showing moderate complete circumferential membrane staining (score 2+) and demonstrating HER2 gene amplification defined as a FISH ratio of HER2 gene copies to chromosome 17 signals of >2.2. or as >5 HER2 gene copies per nucleus in CISH analysis.

Patients with a negative or equivocal overall result (FISH test ratio of <2.2, <6.0 HER2 gene copies per nucleus) and staining scores of 0,1+, 2+ or 3+ (in 30% or less neoplastic cells) by IHC are not eligible for participation in the trial.

* Age ≥18
* Eastern Cooperative Oncology Group (ECOG) performance status ≤1 (Appendix B)
* Adequate bone marrow function (ANC >1.0 x 109/l, platelets >100 x 109/l)
* Adequate hepatic function (ALAT, ASAT and bilirubin <2 times upper limit of normal)
* Adequate renal function (creatinine clearance >60 ml/min)
* LVEF ≥50% measured by echocardiography or MUGA
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Signed written informed consent

Exclusion Criteria:

* No previous radiation therapy or chemotherapy
* No other malignancy except carcinoma in situ, unless the other malignancy was treated ≥5 years ago with curative intent without the use of chemotherapy or radiation therapy.
* No current pregnancy or breastfeeding. Women of childbearing potential must use adequate contraceptive protection.
* No evidence of distant metastases. Staging examinations must have included a chest radiograph, an ultrasound examination of the liver and an isotope bone scan. Abnormal uptake on the isotope bone scan can only be accepted if MRI, CT-scan, or plain radiograph excludes bone metastases.
* No concurrent anti-cancer treatment or another investigational drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2008-09; Primary Completion 2011-08 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Pathologic complete response (pCR) rate at surgery | at the completion of neo-adjuvant chemotherapy

SECONDARY OUTCOMES:
To describe disease-free and overall survival | during routine follow up visits after surgery

CONTACTS AND LOCATIONS:
Overall Officials: G S Sonke, MD, Principal Investigator — NKI-AvL
Locations (9):
- Netherlands (9):
  - Medisch Centrum Alkmaar, Alkmaar
  - NKI-AVL, Amsterdam
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Reinier de Graaf Gasthuis, Delft
  - Catharina Ziekenhuis, Eindhoven
  - Kennemer Gasthuis, Haarlem
  - Leids Universitair Medisch centrum, Leiden
  - Medisch Centrum Haaglanden, Leidschendam
  - Sint Antonius Ziekenhuis, Nieuwegein